CLINICAL TRIAL: NCT03128255
Title: I-124 PET/US for Benign Thyroid Diseases - Blinded, Multicentric Assessment of Augmented Thyroid Work-up Versus Regular Thyroid Diagnostics
Brief Title: Fusion UltraSound Imaging Of the Thyroid GlaNd With I-124 PET. Evaluation of Nodule Allocation.
Acronym: FUSION iENA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: I-124-04/2017
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Nodule; Thyroid Diseases; Thyroid Goitre
Keywords: Fusion; Hybrid Imaging; Mapping; Iodine; Ultrasound
MeSH Terms: conditions — Thyroid Nodule; Thyroid Diseases; Goiter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Thyroid Work-up: Nuclear Medicine physicians evaluate up to 34 cases of patients who have received regular thyroid diagnostics. Data and images of patient characteristics, laboratory results, ultrasonography loops and planar 99mTcO4 scintigraphy are provided and the physicians are asked to assign the function (hypo-, iso-, hyperfunctional) to predefined thyroid nodules visible on ultrasonography.
- Regular Thyroid Work-up and I-124 PET/US: Nuclear Medicine physicians evaluate up to 34 cases of patients who have received regular thyroid diagnostics and additional I-124 PET/CT, followed by I-124 PET/US (administration of I-124 was not subject of this study). Data and images of patient characteristics, laboratory results, ultrasonography loops, planar 99mTcO4 scintigraphy as well as I-124 PET/US loops are provided and the physicians are asked to assign the function (hypo-, iso-, hyperfunctional) to predefined thyroid nodules visible on ultrasonography.
  Interventions: Other: Assessment of already preacquired I-124 PET/US

INTERVENTIONS:
Other: Assessment of already preacquired I-124 PET/US — Assessment of preacquired I-124 PET/US by review of anonymous digital case files
  Groups: Regular Thyroid Work-up and I-124 PET/US

SUMMARY:
Regular thyroid diagnostics versus augmented thyroid work-up with additional I-124 PET/US fusion for metabolic-sonographic nodule allocation in patients with benign thyroid diseases

ELIGIBILITY:
Inclusion Criteria:

* patients with thyroidal nodules,
* euthyroidism
* Uptake >0,5% on Tc-99m-pertechnetate- scintigraphy

Exclusion Criteria:

* thyroid medications in the last 6 months
* Iodine exposition in the last 6 months
* thyroid surgery or radioiodine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of patients with unclear findings on regular thyroid work-up who had received additional I-124-PET/US in our institution.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Metabolic-sonographic nodule allocation | 1 year
  The number of correct assignments of metabolic function of each nodule will be assessed for each group seperately. A three-point scale will be used for evaluation of the nodule's function and the degree of the physicians certainty will be investigated using a four-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No